CLINICAL TRIAL: NCT03960528
Title: Investigation of Erector Spinae Plane Block Effect in Spine Surgery
Brief Title: The Effect of Erector Spinae Plane Block Performed Under Direct Vision on Postoperative Pain in Spine Surgery
Acronym: ESPOUSES
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bezmialem Vakif University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: S003
Record Dates: First submitted 2019-05-21; First posted 2019-05-23 (Actual); Last update posted 2021-09-08 (Actual); Status verified 2021-09

CONDITIONS: Acute Pain
Keywords: spine surgery; postoperative pain; perioperative analgesia; postoperative opioid requirement
MeSH Terms: conditions — Acute Pain; Pain, Postoperative | interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Under direct vision erector spinae plane block (Active Comparator): 20 ml bupivacaine 0,25%+ lidocaine 1% used for the infiltration between the transverse process and the erector spinal muscle under direct vision on each side.
  Participants will receive morphine iv PCA in the postanesthesia care unit( 0.5mg / ml 2cc bolus 8 min lock time 2cc/h infusion)
  Interventions: Procedure: Erector spinae plane block
- Control group (Sham Comparator): 20 ml NaCl 0,9% used for the infiltration between the transverse process and the erector spinal muscle under direct vision on each side.
  Participants will receive morphine iv PCA in the postanesthesia care unit( 0.5mg / ml 2cc bolus 8 min lock time 2cc/h infusion)
  Interventions: Procedure: Control group

INTERVENTIONS:
Procedure: Erector spinae plane block — Bilateral 20 ml Bupivacaine 0.25% + lidocaine 1% injected between erector spinae muscles and transverse process under direct vision.
  Other Names: ESP block
  Arms: Under direct vision erector spinae plane block
Procedure: Control group — 20 ml NaCl 0,9% used for the infiltration between the transverse process and the erector spinal muscle under direct vision on each side.
  Other Names: Sham comparator
  Arms: Control group

SUMMARY:
Spine surgery is typically associated with severe postoperative pain. Although the number of spine surgeries has increased day by day, postoperative pain management have been limited. The recently described erector spinae plane block (ESPB) is obtained by applying the local anesthetic drug between the fascia of the erector spinae muscles and the transverse process of the vertebrae. Anatomical and radiological investigations in fresh cadavers suggest that the potential place of influence of ESPB is dorsal and ventral spinal nerve roots. A small number of publications showing the analgesic efficacy of ESP in spinal surgery have been reported in the literature. The erector spinae muscles are easily identified during spine surgery, and erector spinae plane blocks can be performed under direct vision rather than via ultrasound guidance or simply using anatomical landmarks. Therefore, the investigators aim to observe the efficacy of the under direct vision erector spinae plane block on pain scores after spinal surgery.

DETAILED DESCRIPTION:
Approval from the university local ethics committee will be obtained. Participans will be informed about the potential benefits and complications after the study protocol has been fully and thoroughly explained. After premedication with 0.03 mg / kg iv midazolam, participans will be noninvasively monitored by taking into the operating room (heart rate, blood pressure, pulse oximetry). Anesthesia induction will delivered with fentanyl 1mcg / kg, propofol 2 mg / kg and rocuronium 0.6 mg / kg. The maintenance of anesthesia will be achieved by infusion of sevoflurane 2-3% in 50% O2/50% medical air and remifentanil infusion of 0.1-0.5 mcg / kg / min. Thirty minutes before end of the surgery, all patients were intravenously administered 1 mg/kg tramadol HCl and 1gr paracetamol.

Under direct vision ESPB technique: Erector spinae muscles and transverse processes will be identified by the surgeon. At the end of the surgery 20 ml bupivacaine 0.25%/lidocaine 1% mixture will be injected to the between of the erector spinae muscles and transverse processes bilaterally. In the sham comparator group, 20 ml of isotonic saline will be administered bilaterally by the surgeon as described above.

After the surgery, 1 g paracetamol was intravenously administered once every 8 h. A patient-controlled analgesia (PCA) device, which was prepared using morphine, was attached to the patients and was programmed to administer concentration 0.5mg / ml ( 2cc bolus 8 min lock time 2cc/h infusion). This administration continued for 24 h. Postoperative pain was assessed using visuel analog scale (VAS) (VAS 0 = no pain, VAS 10 = most severe pain ). Duration at postanesthesia care unit (PACU) was recorded right from 0 h. VAS scores at 0, 1, 6, 12 and 24 h were recorded. Postoperative nausea and vomiting (PONV) was evaluated using a numeric ranking scale (0 = no PONV, 1 = mild nausea, 2 = severe nausea or vomiting once attack, and 3 = vomiting more than once attack). If PONV score was >2, the antiemetic metoclopramide Hcl 10mg was intravenously administered.

ELIGIBILITY:
Inclusion Criteria:

1. 20-75 years
2. ASA 1-2-3
3. Patients scheduled for elective surgery

Exclusion Criteria:

1. Patients with previous neurological disease symptoms (TIA, syncope, dementia, etc.)
2. Allergy to drugs
3. Major cardiac disease
4. Renal failure
5. Psychiatric disease
6. Patients who refuse to participate in the study
7. Chronic back and lower back pain
8. Body mass index <18.5 and >40

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2019-04-18 (Actual); Primary Completion 2020-01-10 (Actual); Study Completion 2020-02-10 (Actual)

PRIMARY OUTCOMES:
Total morphine consumption | 1 day
  The total amount of morphine given by patient controlled analgesia in 24 hours will be recorded

SECONDARY OUTCOMES:
Pain intensity score | 1 day
  Changes in Numeric Rating Scale (NRS) will be recorded at postoperative 1, 6, 12, 24 hour. The NRS is a segmented numeric version of the visual analog scale (VAS) in which a respondent selects a whole number (0-10 integers) that best reflects the intensity of patient pain. Each item is scored 0-10( 0:no pain 10: pain as bad as can be )
Postoperative nausea and vomiting | 1 day
  Changes in Numeric Rank Score will be recorded at postoperative 1, 6, 12, 24 hour. Numeric rank score 0-3(0: no nausea and vomiting; 1:have nausea, no vomiting; 2:once vomiting attack; 3: have two or more vomiting attacks)

CONTACTS AND LOCATIONS:
Overall Officials: Serdar YEŞİLTAŞ, Instructor, Principal Investigator — BEZMİALEM VAKIF UNIVERSITY
Locations (1):
- Bezmialem Vakıf University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No